CLINICAL TRIAL: NCT02694965
Title: Understanding Immunotherapy Resistance Mechanisms in Advanced Melanoma
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00059349
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2023-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Low risk biopsy and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stage IV/Unresectable Stage III Melanoma: Observational - Eligible patients with stage IV/unresectable stage III melanoma selected to undergo treatment with an anti-CTLA-4 antibody, an anti-PD-1 antibody, an anti-PD-L1 antibody, or a combination of an anti-CTLA-4 antibody/anti-PD-1 antibody will be asked to participate in the study by the Principal Investigator, co-Investigators, or clinical staff.
  Interventions: Other: observational
- Stage III/IV Adjuvant Melanoma: Observational - 1) Patients either undergoing resection of stage III or stage IV melanoma or have previously undergone resection and who are considered candidates for adjuvant anti-PD-1 antibody immunotherapy. 2) Patients who previously underwent resection of stage III or stage IV melanoma and received prior adjuvant anti-PD-1 antibody immunotherapy and have subsequently developed recurrent melanoma.
  Interventions: Other: observational

INTERVENTIONS:
Other: observational

SUMMARY:
Purpose of the study:

The investigators are proposing that melanomas which respond and develop eventual disease stability in response to checkpoint inhibitor immunotherapy undergo a genetic program promoting secondary resistance.

DETAILED DESCRIPTION:
Understanding these genetic alterations and the factors which contribute to this process would be critical for the identification of novel immunotherapeutic targets which may synergize with the T cell-targeted checkpoint inhibitors. Furthermore, this work promises to provide greater insight into tumor-mediated immune evasion mechanisms and primary immunotherapy resistance, potentially unveiling predictive markers of clinical response for our expanding arsenal of immune checkpoint inhibitor therapies.

Many patients who exhibit a response to the anti-PD-1 antibodies develop a prolonged course of disease stability which resembles the equilibrium phase of the previously proposed process of cancer immunoediting. This state of equipoise has been hypothesized to involve genetic alterations that promote immune evasion and, in some cases, lead to the development of tumor escape. Based on our data, the investigators propose that melanomas that develop a period of disease stability in response to anti-PD-1 immunotherapy exhibit genetic alterations that suppress the effectiveness of anti-tumor immunity. Our previous studies indicate that the tumor-derived factors that play a role in the paracrine signaling pathways capable of regulating nearby stromal cell populations are more likely to be critical immune regulators of the tumor microenvironment. Therefore, the investigators will focus our studies on those differentially expressed genes which encode soluble proteins using an available prediction algorithm. Those genes identified by this study to be differentially expressed in the melanoma tissues of patients demonstrating a clinical response to immune checkpoint inhibitor therapy will be further evaluated in transgenic autochthonous melanoma models.

ELIGIBILITY:
Arm 1 Subject Selection:

Eligible patients with stage IV/unresectable stage III melanoma selected to undergo treatment with an anti-CTLA-4 antibody, an anti-PD-1 antibody, an anti-PD-L1 antibody, or a combination of an anti-CTLA-4 antibody/anti-PD-1 antibody will be asked to participate in the study by the Principal Investigator, co-Investigators, or clinical staff.

Inclusion Criteria

* Patients with stage III or IV melanoma, with melanoma validated by histology or cytology
* Patients may participate with primary cutaneous melanomas of unknown primary site
* Age ≥ 18 years
* ECOG performance status of 0-2
* Life expectancy of at least 6 months
* Patients with active disease will be treated with either an anti-CTLA-4 antibody , an anti-PD-1 antibody, an anti-PD-L1 antibody, or a combination of an anti-CTLA-4 antibody/anti-PD-1 antibody (combined therapy regimens with any other agents are not allowed on this study).
* Patient must have a measurable systemic lesion defined as greater than or equal to 10 mm based on PET CT/CT/MRI imaging. Pretreatment PET CT/CT imaging must be performed ≤ 42 days prior to treatment initiation ).
* Patients with target skin lesions must equal at least 10 mm when their longest diameters are aggregated. Target skin lesions (5 maximum) must be at least 5 mm in their longest diameter to be considered measurable by caliper or ruler
* Those patients with a failed biopsy attempt or those with disease that is not amenable to biopsy will still be eligible for enrollment and will only undergo blood draws during the study protocol.
* Both men and women of all races and ethnic groups are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document
* Patients with intra-cranial disease or disease involving the central nervous system are eligible

Exclusion Criteria

* Patients with a history of a systemic autoimmune disease (eg systemic lupus erythematosus) requiring active therapy
* Patients with a history of another malignancy within the last 5 years except for those patients felt by the treating physician to be cured of that malignancy
* Patients with a diagnosis of a mucosal or ocular melanoma
* Patients who have undergone adjuvant locoregional radiation therapy if less than 4 weeks prior to day of initial biopsy
* Patients who have had prior cytotoxic chemotherapy if less than 6 weeks prior to day of initial biopsy
* Patients who have had prior interferon therapy if less than 4 weeks prior to day of initial biopsy
* Patients who have had prior anti-CTLA-4 antibody or anti-PD-1 antibody or anti-PD-L1 antibody therapy if less than 4 weeks prior to day of initial biopsy
* Patients who have had prior IL-2 therapy if less than 4 weeks prior to day of initial biopsy
* Patients who have had prior BRAF inhibitor and/or MEK inhibitor therapy if less than 4 weeks prior to day of initial biopsy
* Patients who have received an immunotherapy agent on a previous clinical trial protocol if less than 4 weeks prior to day of initial biopsy
* Patients who are undergoing active steroid therapy if the dose exceeds physiologic steroid doses (equivalent of prednisone 10 mg po daily or less)
* Patients with ongoing or active infection
* Pregnant patients
* Patients with any laboratory test values or serious pre-existing medical condition, that in the opinion of the investigator, makes the patient unsuitable for the study
* Patients unable to comply with the requirements of the study protocol

Arm 2 Subject Selection:

The following patients will be asked to participate in the study by the Principal Investigator, co-Investigators, or clinical staff: 1) Patients either undergoing resection of stage III or stage IV melanoma or have previously undergone resection and who are considered candidates for adjuvant anti-PD-1 antibody immunotherapy. 2) Patients who previously underwent resection of stage III or stage IV melanoma and received prior adjuvant anti-PD-1 antibody immunotherapy and have subsequently developed recurrent melanoma.

Inclusion Criteria

* Patients with a current diagnosis of stage III or IV melanoma or a history of stage III or IV melanoma, with melanoma validated by histology or cytology
* Age ≥ 18 years
* ECOG performance status of 0-2
* Patients selected for future adjuvant anti-PD-1 antibody immunotherapy following resection of stage III or stage IV melanoma or patients who received prior adjuvant anti-PD-1 antibody immunotherapy for stage III or IV melanoma and have developed recurrent disease based on physical exam and/or CT/PET CT cross-sectional imaging
* Those patients with a failed biopsy attempt or those with disease that is not amenable to biopsy will still be eligible for enrollment and will only undergo blood draws during the study protocol. Of note, any tissue subjected to prior adjuvant radiation therapy will not be considered for further tissue sampling on this protocol.
* Both men and women of all races and ethnic groups are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document
* Patients with intra-cranial disease or disease involving the central nervous system are eligible

Exclusion Criteria

* Patients with a history of a systemic autoimmune disease (eg systemic lupus erythematosus) requiring active therapy
* Patients with a history of another malignancy within the last 5 years except for those patients felt by the treating physician to be cured of that malignancy
* Patients with a diagnosis of a mucosal or ocular melanoma
* Patients who have had prior cytotoxic chemotherapy if less than 6 weeks prior to day of initial biopsy
* Patients who have undergone adjuvant locoregional radiation therapy if less than 4 weeks prior to day of initial biopsy
* Patients who have had prior interferon therapy if less than 4 weeks prior to day of initial biopsy
* Patients who have had prior anti-CTLA-4 antibody or anti-PD-1 antibody or anti-PD-L1 antibody therapy if less than 4 weeks prior to day of initial biopsy
* Patients who have had prior IL-2 therapy if less than 4 weeks prior to day of initial biopsy
* Patients who have had prior BRAF inhibitor and/or MEK inhibitor therapy if less than 4 weeks prior to day of initial biopsy
* Patients who have received an immunotherapy agent on a previous clinical trial protocol if less than 4 weeks prior to day of initial biopsy
* Patients who are undergoing active steroid therapy if the dose exceeds physiologic steroid doses (equivalent of prednisone 10 mg po daily or less)
* Patients with ongoing or active infection
* Pregnant patients
* Patients with any laboratory test values or serious pre-existing medical condition, that in the opinion of the investigator, makes the patient unsuitable for the study
* Patients unable to comply with the requirements of the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Arm 1:
  Eligible patients with stage IV/unresectable stage III melanoma selected to undergo treatment with an anti-CTLA-4 antibody, an anti-PD-1 antibody, an anti-PD-L1 antibody, or a combination of an anti-CTLA-4 antibody/anti-PD-1 antibody will be asked to participate in the study by the Principal Investigator, co-Investigators, or clinical staff.
  Arm 2:
  1) Patients either undergoing resection of stage III or stage IV melanoma or have previously undergone resection and who are considered candidates for adjuvant anti-PD-1 antibody immunotherapy. 2) Patients who previously underwent resection of stage III or stage IV melanoma and received prior adjuvant anti-PD-1 antibody immunotherapy and have subsequently developed recurrent melanoma.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2016-01; Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Observational - Correlate changes in gene expression upon disease progression or recurrence | up to 3 years
  Arm 1: Differential gene expression will be compared in samples from pre-treatment and disease progression.
  Arm 2: Differential gene expression will be compared in samples from pre-treatment and disease recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Hanks, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided